CLINICAL TRIAL: NCT01564732
Title: Multicenter Prospective Randomized Clinical Trial of Plicated Laparoscopic Adjustable Gastric Banding
Brief Title: Multicenter Prospective Randomized Controlled Trial of Plicated Laparoscopic Adjustable Gastric Banding
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor withdrew funding.
Sponsor: Dana Portenier, MD (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor-Investigator, Dana Portenier, MD, Assistant Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00033638
Record Dates: First submitted 2012-03-07; First posted 2012-03-28 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; gastric band
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard-LAGB (Active Comparator): Subjects will be blinded and randomly assigned to the Standard Laparoscopic Gastric Banding(SLAGB)arm of the study. These subjects will receive the standard of care or standard laparoscopic gastric banding surgery.Subjects will be followed for a period of approximately 36 months.
  Interventions: Device: Standard-LAGB
- Plicated-LAGB (Experimental): Subjects will be blinded and randomly assigned to the Plicated Laparoscopic Gastric Banding(PLAGB)arm of the study. These subjects will receive the plicated laparoscopic gastric banding surgery with involves the placement of plication sutures to "anchor" the redundant stomach around the newly placed device. Subjects will be followed for a period of approximately 36 months.
  Interventions: Device: Plicated-LAGB

INTERVENTIONS:
Device: Standard-LAGB — The laparoscopic adjustable gastric banding (LAGB) procedure is a safe, effective, and durable treatment option for refractory morbid obesity and its related health consequences.5 This minimally invasive technique is now a popular approach for bariatric surgery, and it offers obvious advantages such as decreased operating time, shorter hospital stay (often same day surgery), and favorable complication rates as compared with other bariatric procedures.
  Other Names: Standard Laparoscopic Adjustable Gastric Banding Surgery
  Arms: Standard-LAGB
Device: Plicated-LAGB — At the time of LAGB placement, plication sutures can be placed along the body & greater curvature of the stomach to "tighten" and "cinch up" the stomach in a sleeve-like orientation. It was recently reported that this modified technique of plicated LAGB could result in lower band slippage complication rates and faster, early weight loss.
  Other Names: Plicated Laparoscopic Adjustable Gastric Banding Surgery
  Arms: Plicated-LAGB

SUMMARY:
The purpose of this study is to compare plicated laparoscopic adjustable gastric banding (PLAGB) to standard laparoscopic adjustable gastric banding (SLAGB) in a prospective randomized clinical trial. We hypothesize the plicated procedure will provide greater short- and long-term excess weight loss than the standard procedure. There exists little prospective randomized data regarding this topic and the recent position statement from the American Society for Metabolic and Bariatric Surgery (ASMBS) encourages this type of study. Further information on background and design of this study are provided in the detailed description.

DETAILED DESCRIPTION:
Morbid obesity is a major problem affecting the lives of millions in the US. As of 2008, overall prevalence of obesity as defined by body mass index (BMI) greater than 30 kg/m2 was 33.8%.1 Obesity adversely affects the lives of millions of Americans by increasing the risk for co-morbid conditions such as diabetes mellitus, obstructive sleep apnea, hypertension, and even certain cancers.2-4 The laparoscopic adjustable gastric banding (LAGB) procedure is a safe, effective, and durable treatment option for refractory morbid obesity and its related health consequences.5 This minimally invasive technique is now a popular approach for bariatric surgery, and it offers obvious advantages such as decreased operating time, shorter hospital stay (often same day surgery), and favorable complication rates as compared with other bariatric procedures.4,5

One of the biggest drawbacks to LAGB [when compared to the 'gold standard' of bariatric surgery: Roux-en-Y gastric bypass] is that patients tend to have a slower, less dramatic weight loss in the first few months after surgery.5-7 In addition, the LAGB procedure is associated with an approximate 3% chance of "band slippage" complications.8 In order to address some of these issues modifications in the technique of LAGB surgery have been made. Techniques such as a "pars-flaccida approach" to tissue dissection and the placement of plication sutures to "anchor" the redundant stomach around the newly placed band device were introduced and shown to have positive results in reducing band complication rates.8 More recently, sleeve gastrostomy procedures (the greater curvature and significant portion of the body of the stomach is resected over a sizing bougie; leaving a narrow 'sleeve' of stomach) have also become popular in treating patients with morbid obesity.9 Combining these concepts, a modified technique of plicated LAGB was introduced.

At the time of LAGB placement, plication sutures can be placed along the body & greater curvature of the stomach to "tighten" and "cinch up" the stomach in a sleeve-like orientation. It was recently reported that this modified technique of plicated LAGB could result in lower band slippage complication rates and faster, early weight loss.8

However, as of today there exists no prospective, randomized study that compares the outcomes of this modified surgical technique to the standard procedure (SLAGB).

This is a prospective randomized clinical trial comparing PLAGB versus SLAGB. All adult (age older than 18 years) morbidly obese patients meeting NIH criteria for bariatric surgery (BMI > 35 + co-morbid disease or BMI > 40) who are undergoing bariatric surgery at the Duke Metabolic and Weight Loss Surgery Center and the University of Pittsburgh Medical Center will be recruited. All enrolled patients will be randomly assigned to either the SLAGB (control) group or the PLAGB (study) group. Variables to be studied include patient age, gender, ethnicity, co-morbid disease conditions, height, weight, BMI, intra-operative data such as operative time and blood loss, and post-operative outcomes including length of hospital stay, complication rates, weight loss, and co-morbid disease resolution. In addition, each patient will complete standardized surveys rating their satisfaction from surgery, their quality of life (OWL-QOL-17), and their sleepiness (Epworth Sleepiness Scale) at three distinct time intervals: pre-operatively and at weeks 24 & 48.

Each subject will be followed and data collected according to the following schedule of visits:

Study Visit Schedule:

Year 1:

Visit 1: Screening Visit Visit 2: Day 0 (surgery) Visit 3: Week 2 (+/- 2 days) Visit 4: Week 4 (1 month) Visit 5: Week 8 (2 months) Visit 6: Week 12 (3 months) Visit 7: Week 16 (4 months) Visit 8: Week 20 (5 months) Visit 9: Week 24 (6 months) Visit 10: Week 30 Visit 11: Week 36 Visit 12: Week 42 Visit 13: Week 48

Year 2:

Visit 14: Week 60 Visit 15: Week 72 Visit 16: Week 84 Visit 17: Week 96

Year 3:

Visit 18: Week 128 (2.5 yrs) Visit 19: Week 156 (3 yrs)

Data gathered from PLAGB subjects will be compared to SLAGB controls. Pre- and post-operative care will be delivered consistent with our established protocols and standard practices; without regard to surgical approach. This includes a standard preoperative evaluation and patient education period followed by surgery. After surgery, patients are usually discharged from the hospital within the first 24 hours. Follow-up of patients will include an initial post-discharge clinic visit within the first 2 weeks, and subsequent visits scheduled at the time intervals as listed above. Subjects will be followed for a period of approximately 12 months.

This study compares a modified bariatric surgical approach. PLAGB will be studied and compared to the SLAGB procedure through a prospective randomized clinical trial.

Please note: Per our FDA approved modification of 6/18/2014, all study specific testing was eliminated, and only safety assessments were completed in the surgical office at 6 months and 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria: Subjects must meet the following criteria to be eligible for study entry:

1. Age between 18-60 years,
2. Morbidly obese:

a. BMI > 40, or b. BMI > 35 + co-morbid obesity related disease condition c)BMI < or equal to 55

Exclusion Criteria: Subjects meeting the following criteria will be excluded from study entry:

1. Patients with any major medical problems contraindicating surgery (eg.myocardial infarct within last 6 months, cancer within last 5 years, end stage renal/liver disease, etc.)
2. Patients with a medically treatable cause of obesity (eg. untreated hypothyroidism, Prader-Willi, etc.)
3. Patients who elect to undergo a surgery other than a PLAGB or SLAGB
4. Patient who is unwilling to be randomized to PLAGB or SLAGB
5. Pregnant or planning pregnancy within 12 months
6. Alcohol or drug addiction
7. Established infection anywhere in the body at the time of surgery
8. Previous history of bariatric surgery, gastric surgery, intestinal obstruction, or adhesive peritonitis.
9. Family or patient history of autoimmune disease
10. Hiatal Hernia > 3cm (as reported per radiology on pre-operative swallow study)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana D Portenier, MD, Principal Investigator — Duke University; Carol McCloskey, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Flegal KM, Carroll MD, Ogden CL, Curtin LR. Prevalence and trends in obesity among US adults, 1999-2008. JAMA. 2010 Jan 20;303(3):235-41. doi: 10.1001/jama.2009.2014. Epub 2010 Jan 13. PMID 20071471
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Pories WJ. Bariatric surgery: risks and rewards. J Clin Endocrinol Metab. 2008 Nov;93(11 Suppl 1):S89-96. doi: 10.1210/jc.2008-1641. PMID 18987275
- [Background] Longitudinal Assessment of Bariatric Surgery (LABS) Consortium; Flum DR, Belle SH, King WC, Wahed AS, Berk P, Chapman W, Pories W, Courcoulas A, McCloskey C, Mitchell J, Patterson E, Pomp A, Staten MA, Yanovski SZ, Thirlby R, Wolfe B. Perioperative safety in the longitudinal assessment of bariatric surgery. N Engl J Med. 2009 Jul 30;361(5):445-54. doi: 10.1056/NEJMoa0901836. PMID 19641201
- [Background] Gravante G, Araco A, Araco F, Delogu D, De Lorenzo A, Cervelli V. Laparoscopic adjustable gastric bandings: a prospective randomized study of 400 operations performed with 2 different devices. Arch Surg. 2007 Oct;142(10):958-61. doi: 10.1001/archsurg.142.10.958. PMID 17938309
- [Background] Cottam DR, Atkinson J, Anderson A, Grace B, Fisher B. A case-controlled matched-pair cohort study of laparoscopic Roux-en-Y gastric bypass and Lap-Band patients in a single US center with three-year follow-up. Obes Surg. 2006 May;16(5):534-40. doi: 10.1381/096089206776944913. PMID 16687018
- [Background] Hussain A, Mahmood H, El-Hasani S. Gastric plication can reduce slippage rate after laparoscopic gastric banding. JSLS. 2010 Apr-Jun;14(2):221-7. doi: 10.4293/108680810X12785289144241. PMID 20932373
- [Background] Lee CM, Cirangle PT, Jossart GH. Vertical gastrectomy for morbid obesity in 216 patients: report of two-year results. Surg Endosc. 2007 Oct;21(10):1810-6. doi: 10.1007/s00464-007-9276-y. Epub 2007 Mar 14. PMID 17356932
- [Background] Lancaster RT, Hutter MM. Bands and bypasses: 30-day morbidity and mortality of bariatric surgical procedures as assessed by prospective, multi-center, risk-adjusted ACS-NSQIP data. Surg Endosc. 2008 Dec;22(12):2554-63. doi: 10.1007/s00464-008-0074-y. Epub 2008 Sep 20. PMID 18806945

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 subjects consented to participate: 1 from Duke University and 16 from the University of Pittsburgh, 6 had not completed surgery before the study termination (2 withdrawn by the PIs and 4 were still in their pre-surgical workup). 11 participants had surgery and were randomized (per the protocol) to plicated band (PLAGB) or standard band (SLAGB).
Period: Overall Study
Arm/Group | Standard-LAGB | Plicated-LAGB
Started | 6 | 5
Completed | 0 | 0
Not Completed | 6 | 5
Not completed — Early termination by the study sponsor | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard-LAGB | Plicated-LAGB | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Customized [Number; unit: participants]
  ≥18 to ≤60 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Time Frame: 36 months
Population: Data not collected.
Arm/Group | Standard-LAGB | Plicated-LAGB
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Quality of Life
Time Frame: 36 months
Population: data not collected
Arm/Group | Standard-LAGB | Plicated-LAGB
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quantitative Change in Hypertension
Description: Systolic and Diastolic Blood Pressure will be measured over the scheduled visits and the change in preoperative and postoperative blood pressure will be determined. We will also assess the need for medications to treat hypertension before and after surgery.
Time Frame: 36 months
Population: Data not collected.
Arm/Group | Standard-LAGB | Plicated-LAGB
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Quantitative Change in Diabetes
Description: Blood Sugar will be measured over the scheduled visits and the change in preoperative and postoperative glucose levels will be determined. We will also assess the need for medications to treat diabetes before and after surgery.
Time Frame: 36 months
Population: Data not collected
Arm/Group | Standard-LAGB | Plicated-LAGB
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Quantitative Change in Hyperlipidemia
Description: Lipid levels will be measured annually for 3 years and the change in preoperative and postoperative levels will be determined. We will also assess the need for medications to treat hyperlipidemia before and after surgery.
Time Frame: 36 months
Population: Data not collected.
Arm/Group | Standard-LAGB | Plicated-LAGB
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Quantitative Change in Hypertriglyceridemia
Description: Triglyceride levels will be measured annually for 3 years and the change in preoperative and postoperative levels will be determined. We will also assess the need for medications to treat hypertriglyceridemia before and after surgery.
Time Frame: 36 months
Population: Data not collected.
Arm/Group | Standard-LAGB | Plicated-LAGB
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Standard-LAGB | Plicated-LAGB
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 1/6 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard-LAGB (N=6) | Plicated-LAGB (N=5)
3mm splenic capsular tear (Surgical and medical procedures) | 0 | 1
Left hand laceration (Injury, poisoning and procedural complications) | 0 | 1
2cm abrasion of the left hepatic lobe (Surgical and medical procedures) | 1 | 0
rotator cuff tear (Injury, poisoning and procedural complications) | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 1
premature atrial contractions (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No